CLINICAL TRIAL: NCT06655922
Title: The Clinical Value of FAPI Imaging in Assessing Chronic Total Occlusion Lesions in Patients with Coronary Heart Disease (FACT Trial)
Brief Title: FAPI Imaging Assessment of Chronic Total Occlusion
Acronym: FACT
Status: Recruiting | Type: Observational
Sponsor: Lin Zhao (Other)
Collaborators: Beijing Chao Yang Hospital (Other)
Responsible Party: Sponsor-Investigator, Lin Zhao, Cheif of Cardiovascular department, Beijing Chao Yang Hospital
Organization: Beijing Chao Yang Hospital (Other)
Other Study IDs: 2024-772-1
Record Dates: First submitted 2024-10-05; First posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Chronic Total Occlusion (CTO)
Keywords: Coronary Heart Disease; Fibroblast activation protein inhibitor; Percutaneous coronary intervention; Imaging; Prognosis
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with at least one untreated CTO at basal angiography: Total occlusion in any major coronary vessel or relevant side branches [reference vessel diameter ≥2.5mm or as judged by two independent interventional cardiologists], with TIMI 0 in the distal segment and at least 3 months old
  Interventions: Diagnostic Test: FAPI Imaging

INTERVENTIONS:
Diagnostic Test: FAPI Imaging — Studies have shown that imaging with radionuclide-labeled fibroblast activation protein inhibitor (FAPI) is a reliable technique for detecting myocardial fibrosis and activated CFs in arteries. Preliminary evidence suggests that FAPI imaging can assess plaque characteristics and the status of myocardial fibrosis in various cardiovascular diseases.

SUMMARY:
This registry will include consecutive patients presenting with at least one chronic total coronary occlusion (CTO) identified via coronary angiography or cardiac computed tomography angiography (CCTA) at our center. Due to the complexity of CTO lesions, both procedural success rates and prognosis improvements are limited. The progression and development of atherosclerotic plaques involve fibroblast activity, contributing to the formation of fibrous caps and calcified nodules through various mechanisms. Myocardial fibrosis within chronically occluded segments is strongly linked to ventricular remodeling and patient prognosis. The activation of cardiac fibroblasts (CFs) is a critical early phase in myocardial fibrosis, playing a key role in fibrotic progression. However, the role of activated CFs in CTO patients has remained unclear, mainly due to the lack of reliable in vivo assessment techniques for detecting CF activation.

Recent studies have demonstrated that radionuclide-labeled fibroblast activation protein inhibitor (FAPI) imaging is an effective and reliable technique for detecting both myocardial fibrosis and activated CFs in arterial plaques. Preliminary data suggest that FAPI imaging can characterize plaque composition and assess the extent of myocardial fibrosis in various cardiovascular conditions. However, its potential to predict the ease of CTO recanalization and subsequent clinical outcomes remains to be fully explored.

The aim of this prospective cohort study is to evaluate the predictive value of FAPI imaging in patients with at least one untreated CTO. All enrolled patients will undergo baseline assessments prior to intervention, including blood tests, clinical evaluations, and imaging studies. These imaging studies will include myocardial FDG/perfusion imaging, FAPI imaging, and resting perfusion imaging. In selected patients, additional evaluations such as stress myocardial perfusion imaging, magnetic resonance imaging (MRI), and echocardiography will also be performed.

For patients undergoing percutaneous coronary intervention (PCI), follow-up assessments will occur at 6 and 12 months. At the 6-month mark, improvements in left ventricular (LV) wall motion will be assessed using resting perfusion imaging. At 12 months, coronary angiography (CAG) will be performed on all patients to evaluate recanalization outcomes. Additionally, myocardial perfusion imaging, magnetic resonance imaging (MRI), and echocardiography may be selectively used to evaluate patients during the 12-month follow-up.

1. To evaluate the ability of FAPI imaging in predicting the difficulty of CTO recanalization.
2. To investigate the role of myocardial FAPI imaging in predicting the improvement of LV wall motion at 6 months, assessed using follow-up single-photon emission computed tomography (SPECT).

By comparing FAPI imaging with conventional prognostic assessment methods, this study aims to clarify the utility of FAPI imaging in both predicting the recanalization complexity and in assessing long-term clinical outcomes in CTO patients.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Presence of at least one untreated CTO at basal angiography (defined as a total occlusion in any major coronary vessel or relevant side branches [reference vessel diameter ≥2.5mm or as judged by two independent interventional cardiologists], with TIMI 0 in the distal segment and at least 3 months old
* Patient has a clinical indication to perform CTO PCI
* Willing to participate and able to understand, read and sign the informed consent document.

Exclusion Criteria:

* Hypersensitivity to aspirin, clopidogrel, or -limus families / or contraindication to antiplatelet agents
* Severe hepatic dysfunction (≥3 times normal reference values)
* Severe chronic kidney disease (estimated Glomerular Filtration Rate [eGFR] <30 mL/min/1.73m2)
* Life expectancy < 1 years
* Pregnant women or women with potential childbearing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting with at least one coronary chronic total occlusion (CTO) on coronary angiogram who will be treated by percutaneous coronary intervention
Sampling Method: Non-Probability Sample
Enrollment: 167 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Improvement of left ventricular (LV) wall motion | 6 months after the procedure
  SPECT images (myocardial perfusion imaging, MPI) were analyzed using QPS/QGS software. Segmental wall motion was semi-quantitatively scored using the American Heart Association (AHA) 17-segment LV model and a five-point scale. 0=normal, 1=mildly hypokinetic, 2=moderately hypokinetic, 3=severely hypokinetic, 4=akinetic, 5=dyskinetic. The improvement of LV wall motion was defined as a decrease of the wall motion score of at least 1 point score.

SECONDARY OUTCOMES:
LV end-systolic volume (ml) | 6 months and 12 months after the procedure
  LV function was assessed by modified Simpson's method.Volumes were obtained by delineation of inner and outer LV contours in end-systolic frames on cardiac SPECT, echocardiography or cardiac magnetic resonance.
LV end-diastolic volume (ml) | 6 months and 12 months after the procedure
  LV function was assessed by modified Simpson's method. LV end-diastolic volume was obtained by delineation of inner and outer LV contours in end-diastolic frames on cardiac SPECT, echocardiography or cardiac magnetic resonance.
LV ejection fraction (%) | 6 months and 12 months after the procedure.
  LV function was assessed by modified Simpson's method. Ejection fraction (EF) was computed from the EDV and ESV as follows:EF=EDV-ESV/EDV on cardiac SPECT, echocardiography or cardiac MRI.
Procedural success | immediately after the procedure.
  Procedural success was defined as successful recanalization of the intended CTO lesion with DES implantation, restoration of Thrombolysis In Myocardial Infarction flow grade 3, and residual diameter stenosis <30% on visual assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Zhao, Ph.D MD, Principal Investigator — Beijing Chaoyang Hospital, Capital Medical University, Beijing, China
Locations (1):
- Beijing Chaoyang Hospital, Capital Medical University, Beijing, China, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Only IPD used in the results publication
Supporting Information: Study Protocol, SAP, ICF
Access Criteria: Need a proposal that describes planned analyses and a data sharing agreement

REFERENCES:
- [Background] Panza JA, Ellis AM, Al-Khalidi HR, Holly TA, Berman DS, Oh JK, Pohost GM, Sopko G, Chrzanowski L, Mark DB, Kukulski T, Favaloro LE, Maurer G, Farsky PS, Tan RS, Asch FM, Velazquez EJ, Rouleau JL, Lee KL, Bonow RO. Myocardial Viability and Long-Term Outcomes in Ischemic Cardiomyopathy. N Engl J Med. 2019 Aug 22;381(8):739-748. doi: 10.1056/NEJMoa1807365. PMID 31433921
- [Background] Perera D, Clayton T, Petrie MC, Greenwood JP, O'Kane PD, Evans R, Sculpher M, Mcdonagh T, Gershlick A, de Belder M, Redwood S, Carr-White G, Marber M; REVIVED investigators. Percutaneous Revascularization for Ischemic Ventricular Dysfunction: Rationale and Design of the REVIVED-BCIS2 Trial: Percutaneous Coronary Intervention for Ischemic Cardiomyopathy. JACC Heart Fail. 2018 Jun;6(6):517-526. doi: 10.1016/j.jchf.2018.01.024. PMID 29852933
- [Background] Wang L, Wang Y, Wang J, Xiao M, Xi XY, Chen BX, Su Y, Zhang Y, Xie B, Dong Z, Zhao S, Yang MF. Myocardial Activity at 18F-FAPI PET/CT and Risk for Sudden Cardiac Death in Hypertrophic Cardiomyopathy. Radiology. 2023 Feb;306(2):e221052. doi: 10.1148/radiol.221052. Epub 2022 Oct 11. PMID 36219116